CLINICAL TRIAL: NCT00809172
Title: Multicenter Randomised Study of Methotrexate Efficacy Versus Cyclosporine in Moderate to Severe Atopic Dermatitis Patients
Brief Title: Study of Methotrexate Efficacy Versus Cyclosporine in Moderate to Severe Atopic Dermatitis Patients
Acronym: METHODA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007.476
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2009-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic-dermatitis; scorad; methotrexate; ciclosporin
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ciclosporin
  Interventions: Drug: Ciclosporin
- 2 (Experimental): Methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Ciclosporin — 5 mg/kg/day per os during 8 weeks after the posology will be changed according to clinical response during the next 16 weeks
  Arms: 1
Drug: Methotrexate — 15 mg/week per os in one tablet during 8 weeks after the posology will be changed according to clinical response during the next 16 weeks
  Arms: 2

SUMMARY:
The systemic treatments for moderate to severe atopic dermatitis (AD) are limited to phototherapy and cyclosporine with the risks respectively of either carcinoma, or hypertension or nephropathy.

Methotrexate was effective in 75% of moderate to severe AD patients with good tolerance in an open retrospective study.

We want to confirm our observations: a non inferiority multicenter clinical trial, methotrexate versus cyclosporine, will be conducted in 100 patients for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years old.
* Both genders eligible for study.
* Moderate to severe AD.
* Scorad > 15.
* Participants must use a contraceptive method during the trial and for 3 months after the end of the trial for female and 5 months for male participants.
* Participants must be able to understand and sign the Informed Consent, and comply with all aspects of the protocol.
* Patients must be registered in a social security system or with a health insurance coverage.

Exclusion Criteria:

* Pregnant or lactating women.
* Evolutive skin disease.
* Patients with a clinically significant disease (chronic, recurrent or active).
* Systemic corticotherapy or immunosuppressive treatment during the previous month, or local corticoid the week before the inclusion.
* Contra-indication to methotrexate and cyclosporine.
* Exposure to phototherapy: cumulative dose > 2000 J/cm2.
* Patients deprived of their civic rights, in custody, or subject to a tutorial, judiciary or administrative decision.
* Patients under a protection measure.
* Patients in a critical medical situation.
* Patients with a personal situation evaluated by the investigator as unable to give optimal participation to the study, or where the study could constitute a risk for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a 50% decrease of scorad ( scorad 50) after 8 weeks of treatment | 36 months

SECONDARY OUTCOMES:
Decrease of scorad by 50% at week4,12,16,20 and 24 | at week4,12,16,20 and 24
Decrease of scorad by 75% and 90 % at week 8 and 24 | at week 8 and 24
quality of life at week 8 and 24 | at week 8 and 24
Concentration of cytokines CCL17 and CCL18 | at week 8 and 24
number of adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Nicolas, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Goujon C, Viguier M, Staumont-Salle D, Bernier C, Guillet G, Lahfa M, Ferrier Le Bouedec MC, Cambazard F, Bottigioli D, Grande S, Dahel K, Berard F, Rabilloud M, Mercier C, Nicolas JF. Methotrexate Versus Cyclosporine in Adults with Moderate-to-Severe Atopic Dermatitis: A Phase III Randomized Noninferiority Trial. J Allergy Clin Immunol Pract. 2018 Mar-Apr;6(2):562-569.e3. doi: 10.1016/j.jaip.2017.07.007. Epub 2017 Sep 28. PMID 28967549